CLINICAL TRIAL: NCT01060436
Title: The Face of Sleepiness
Brief Title: Face of Sleepiness
Acronym: Face
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Ronald D. Chervin, M.D., M.S., Professor of Neurology and Michael S Aldrich Sleep Collegiate Professor of Sleep Medicine, University of Michigan
Other Study IDs: HUM00028854
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2014-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea; sleep disordered breathing; CPAP; BiPAP; treatment outcomes
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CPAP or BiPAP machines — Nightly use of CPAP or BiPAP at a pressure recommended by the subject's treating physician

SUMMARY:
The purpose of this pilot study is to find out whether successful treatment of obstructive sleep apnea makes people look less sleepy, for example by reducing swelling or dark circles under the eyes. In addition, this study will help determine whether facial photographs may be used to help identify patients who should be tested for sleep apnea and daytime sleepiness.

DETAILED DESCRIPTION:
The main symptom of nocturnal sleep disorders is often excessive daytime sleepiness. Although sleepiness can be a major contributor to decreased quality of life, and even mortality, patients frequently grow habituated to their sleepiness, ignoring it and any underlying disorder. One scarcely explored potential consequence that could motivate patients to address sleep disorders is a sleepy facial appearance. No peer-reviewed literature, to our knowledge, has explored whether inadequate or insufficient sleep actually causes changes facial appearance. No published literature has examined the extent to which treatment for sleep disorders might improve such facial changes, and perhaps motivate patients to treat their sleep disorders.

To address these questions in a preliminary manner, therefore, the investigators propose to use cutting-edge photographic technology to assess subtle changes in facial appearance. The investigators will recruit 20 sleepy adult patients who are diagnosed with obstructive sleep apnea, an ideal disease model in which subjects can be tested before and after alleviation of severe sleepiness by home use of continuous positive airway pressure. Results of this pilot study could show for the first time that successful treatment of a chronic sleep disorder improves facial features commonly perceived as an undesirable sign of sleepiness.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18-65
* Recently diagnosed with obstructive sleep apnea, confirmed by polysomnography (sleep study)
* Experiencing daytime sleepiness, based on Epworth Sleepiness Scale
* Scheduled for a positive airway pressure (PAP) titration study (CPAP or BiPAP)
* Willing to use CPAP or BiPAP at pressures prescribed by the treating physician
* Willing to have facial photographs taken before treatment and 2-4 months after nightly use of CPAP or BiPAP

Exclusion Criteria:

* Diagnosed with other sleep, medical or psychiatric disorders that might limit the effectiveness of PAP treatment (such as morbid obesity, emphysema, and neurodegenerative disorders)
* Conditions that may cause daytime sleepiness (such as narcolepsy, primary insomnia, seizure disorders, or major depression)
* Use of medications or herbal remedies that affect sleep and behavior
* History of facial plastic or reconstructive surgery or Botox injections or plans to undergo these types of treatments prior to completing the second study visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University of Michigan Sleep Disorders Clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Photographic assessment of changes in facial indicators of sleepiness (ptosis, flattening or darkening of the external infraorbital surface) after PAP-treatment | 2-4 months after successful nightly use of CPAP or BiPAP

SECONDARY OUTCOMES:
Blinded raters provide visual assessment of relative improvement in facial images of subjects after successful PAP treatment | 2-4 months after successful nightly use of CPAP or BiPAP

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Chervin, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Sleep Disorders Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Chervin RD, Ruzicka DL, Vahabzadeh A, Burns MC, Burns JW, Buchman SR. The face of sleepiness: improvement in appearance after treatment of sleep apnea. J Clin Sleep Med. 2013 Sep 15;9(9):845-52. doi: 10.5664/jcsm.2976. PMID 23997695